CLINICAL TRIAL: NCT00846157
Title: R-CHOP Therapy Compared With R-CHOP Plus Biocell Natural Killer Mixture in Patients With DLBCL (Diffuse Large B Cell Lymphoma);A Randomized, Open-label,Multi-center Trail
Brief Title: Biocell Natural Killer Mixture in Diffuse Large B Cell Lymphoma (DLBCL) Patients
Acronym: NKCell
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: NKBio Co.Ltd. (Industry)
Responsible Party: Lee,Jae-Kyu, Bio Bisiness Headquater/Assistant Manager in Cell Manufacture Team
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NKMGI 4-06
Record Dates: First submitted 2009-02-15; First posted 2009-02-18 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2009-02

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: natural killer cell; DLBCL (Diffuse Large B Cell Lymphoma)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Dendritic Cell Sarcoma, Interdigitating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): Rituximab 375mg/m2 IV administered on day 1. Cyclophosphamide 750mg/m2 IV for 2hours,Adriamycin 50mg/m2 ,Vincristine 1.4mg/m2 IV respectively. Prednisone 60mg P.O. per day for 5 days.
- Active (Active Comparator): R-CHOP plus Natural Killer Cell therapy
  Interventions: Biological: NKM injection

INTERVENTIONS:
Biological: NKM injection — NKCell about 100mg IV for 6times in each chemotherapy period.
  Other Names: NKCell
  Arms: Active

SUMMARY:
Primary objective:

* To compare the event free survival for 3years of R-CHOP plus Biocell Natural Killer Cell to R-CHOP therapy with DLBCL patients.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women of the age between 20 and 70
2. The patients who have measurable lesion using radiograph and have not received chemotherapy and radiation therapy after confirming DCBCL.
3. The patients with Ann arbor Ⅰ, Ⅱ, Ⅲ, Ⅳ
4. The patients who have not received NK / T-Cell lymphocyte therapy.
5. The patients who are expected to survive for at least 3 months.
6. The patients who or whose representative voluntary have written informed consent before performance of any study-related procedure.
7. Women of child bearing potential must have a negative pregnancy test within 7 days prior to study registration and agree to use adequate birth control during study treatment.
8. The patients with ADL classification (ECOG) scale 0, 1, 2
9. Patients who satisfy following hematologic criteria

   * WBC ≥ 3,000 / ㎕
   * platelet count ≥ 75,000 / ㎕
   * serum total bilirubin ≤ two times of upper limit of normal values of each laboratory
   * serum creatinine ≤ two times of upper limit of normal values of each laboratory
10. lymphoma patients who satisfy the following criteria

    * good renal function (GFR> 50)
    * good hepatic function (total bilirubin level ≤ three times of upper limit of normal values of each test laboratory transaminases ≤ 5 times of the upper limit of normal value of each testing laboratory)
11. The patients with negative HIV surface antigen
12. The patients with negative HBV
13. The patients with negative HCV
14. The patients who have not received immunotherapy.
15. The patients who have not experienced tuberculosis infection within recent 6 months.

Exclusion Criteria:

1. The minors under 20 years of age (In accordance with Civil Code)
2. The patients diagnosed with other types of lymphoma
3. The patients who have central nervous system or meningeal involvement by lymphoma.
4. The patients who have contraindication of chemotherapy regimen
5. The patients with another active severe disease.
6. The patients who have history of cancer within 5 years
7. Uncontrolled hypertension patients
8. The patients who have hypersensitivity to Erythropoietin.
9. The patients who have the following diseases or the experience to have following disease within 3 months.

   * Myocardial infarction
   * Unstable coronary disease
   * Uncontrolled cardiac insufficiency.
   * Venous thrombosis
   * Pulmonary embolism
10. The patients who have experience to be treated with the pharmaceutical for clinical trials.
11. Pregnant and lactating women or women of childbearing age not using adequate contraceptive method.
12. The patients with clinically serious bacterial, viral or fungal infection
13. The patients of the test group who have the problem in NK cell cultures (Investigator will decide on this criteria with basis generated during NK cell culture)
14. Patients with autoimmune diseases
15. The patients who underwent visceral resection related with Lymphoma.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2007-09; Primary Completion 2011-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Event Free survival | 3 years

SECONDARY OUTCOMES:
Progression free survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Seok-Goo Cho, MD,PhD, Principal Investigator — Catholic Hematopoietic Stem Cell Transplantation Center in The Catholic University of Korea
Locations (1):
- The Catholic University of korea, Banpo-dong, Seoul, South Korea